CLINICAL TRIAL: NCT04789941
Title: Phase II Trial To Evaluate The Efficiency And Safety Of Neoadjuvant Chemotherapy In Locally Advanced Cancer Cervix
Brief Title: How To Evaluate The Efficiency And Safety Of Neoadjuvant Chemotherapy In Locally Advanced Cancer Cervix
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAI MOHAMED HEMMAT ABDELFATAH ABDELGELIL, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treatment Of Cancer Cervix
Record Dates: First submitted 2020-11-28; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Locally Advanced Cervical Carcinoma
MeSH Terms: interventions — Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm of patients with locally advanced cancer cervix (Experimental): Single arm study to assess the efficacy and safety of use of neoadjuvant cisplatin and irinotecan in treatment of patients with locally advanced cancer cervix.
  A combined regimen of intravenous infusion of cisplatin 80mg/m2 on day 1 with irinotecan 60mg/m2 on day 1 and day 8 of every 21- day cycle for 3 cycles.
  Then, MRI pelvis will be used for assessment of disease response. According to RECIST criteria, patients who will develop at least stable disease, will be sent for radical hysterectomy. Afterwards, 6 weeks after the surgery, another 3 cycles of the same regimen will be given to the participants as adjuvant treatment.
  Interventions: Drug: Cis Platinum + Irinotecan

INTERVENTIONS:
Drug: Cis Platinum + Irinotecan — Studying the efficacy and safety of neoadjuvant cisplatin and irinotecan use in treatment of locally advanced cancer cervix.
  Other Names: No other interventions, investigators are trying only one intervention to test if it could be an alternative effective line for treating the patients with locally advanced cancer cervix.

SUMMARY:
1. This strategy might suggest a therapeutic option to preserve ovarian function in young patients among which locally advanced cancer cervix is common. Based on previous studies, neoadjuvant irinotecan and cisplatin followed by radical hysterectomy and adjuvant chemotherapy has the potential to improve the prognosis compared the concurrent chemo-radiotherapy(CCRT).
2. To offer an alternative effective treatment line replacing concurrent chemo-radiotherapy to avoid dramatic radiotherapy induced complications which might impede a safe successful surgery.

2- To reduce the proportion of patients who will go for radiotherapy, consequently those patients will still have a chance of probable less complicated surgery in case of local recurrence.

3- This study will involve neo-adjuvant chemotherapy (NACT) in treating patients with stage II-III cervical cancer for reducing tumor size, minimizing blood loss during surgery and eradication of possible micro-metastasis.

4- To Improve the likelihood of achieving complete tumor resection after NACT. 5- Investigators will further follow-up those patients for more detailed assessments to confirm whether NACT can improve patients' prognoses, survival, quality of life, and the standard of care.

DETAILED DESCRIPTION:
Treatments for locally advanced cervical cancer, defined as International Federation of Gynecology and Obstetrics (FIGO) stage Ib2-III include primary surgery, neoadjuvant chemotherapy and concurrent chemo-radiotherapy (CCRT). In many countries, CCRT is accepted as the standard therapy for such tumors. However, each of these therapies has both advantages and disadvantages, however, more recently it has been given using neoadjuvant chemotherapy with intravenous irinotecan hydrochloride (CPT-11) and cisplatin. DNA topoisomerases are enzymes that regulate and control DNA topology. Topoisomerase 1 catalyzes the transient cutting of a single DNA strand, the passage of another DNA strand through the break and then resealing of the DNA break. Camptothecin (CPT), an antitumor alkaloid isolated from Camptotheca acuminata, interferes with DNA topoisomerase 1 function. Cisplatin (cis-dichlorodiammineplatinums II) is a first generation platinum compound. Platinum-based NACT followed by radical hysterectomy has been proposed as an alternative approach to radiotherapy or CCRT in locally advanced cervical cancer, especially of squamous cell histology, with objective response rates ranging from 69.4% to 90.2%, pathological optimal response rates ranging from 21.3% to 48.3%, 5-year disease free survival (DFS) rates ranging from 55.4% to 71% and 5-year overall survival(OS) rates ranging from 58.9% to 81%, respectively.

ELIGIBILITY:
Inclusion Criteria:

1 - Patients with histologically confirmed invasive squamous cell carcinoma of the uterine cervix; (ii) FIGO stage system (2018 version): stage II-III 2- No previous treatment. 3- patients with age of 20-75 years at enrollment. 4- Eastern Cooperative Oncology Group performance status (PS) of 0 or 1. 5- Preserved function of major organs (bone marrow, heart, liver and kidney) 6- Lab values within specified ranges, including a neutrophil count greater than 2000/μL, a platelet count greater than 100 000/ mm3 , a hemoglobin level greater than 9.0 g/dL (values after blood transfusion are accepted), levels of aspartate aminotransferase and alanine aminotransferase less than 100 IU/L, a total bilirubin level less than 1.5 mg/dL, a serum creatinine level less than 1.5 mg/dL, creatinine clearance greater than 60 mL/ min.

Exclusion Criteria: :

1. Distinct evidence of infectious disease.
2. Serious concurrent disease (cardiac disease, uncontrolled diabetes mellitus, malignant hypertension and a bleeding tendency).
3. Pregnant women, or women who want to become pregnant.
4. History of serious drug hypersensitivity or drug allergy.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be on cancer cervix patients
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Respectability of the tumor | Evaluation will be done by MRI pelvis after 3 cycles( of the 21- day cycle) of chemotherapy
  Evaluation of the effect of use of neoadjuvant cisplatin and irinotecan on the tumor size when assessed by MRI pelvis cancer
  Evaluation of the tumor size by MRI pelvis after giving 3 cycles of cisplatin and irinotecan. So, baseline( prechemotherapy) MRI pelvis and another re-evaluation MRI pelvis will be used for proper assessment.

SECONDARY OUTCOMES:
2- year relapse free survival(RFS) | 2 years
  Evaluation of the effect of use of neoadjuvant cisplatin and irinotecan on the 2- year RFS of patients with locally advanced cancer cervix
2- year overall survival(OS) | 2 years
  Evaluation of the effect of use of neoadjuvant cisplatin and irinotecan on the 2- year OS of patients with locally advanced cancer cervix
Toxicity profile | 2 years
  Investigators will assess the incidence of treatment related adverse events ( e.g neutropenia,mucositis,renal insufficiency, neuropathy, nausea and vomiting)and its severity on the CTCAE scale of 5 grades ( mild,moderate,severe,life- threatening, and death related to AE. )

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prat J; FIGO Committee on Gynecologic Oncology. Staging classification for cancer of the ovary, fallopian tube, and peritoneum. Int J Gynaecol Obstet. 2014 Jan;124(1):1-5. doi: 10.1016/j.ijgo.2013.10.001. Epub 2013 Oct 22. No abstract available. PMID 24219974
- [Background] Katsumata N, Yoshikawa H, Kobayashi H, Saito T, Kuzuya K, Nakanishi T, Yasugi T, Yaegashi N, Yokota H, Kodama S, Mizunoe T, Hiura M, Kasamatsu T, Shibata T, Kamura T; Japan Clinical Oncology Group. Phase III randomised controlled trial of neoadjuvant chemotherapy plus radical surgery vs radical surgery alone for stages IB2, IIA2, and IIB cervical cancer: a Japan Clinical Oncology Group trial (JCOG 0102). Br J Cancer. 2013 May 28;108(10):1957-63. doi: 10.1038/bjc.2013.179. Epub 2013 May 2. PMID 23640393
- [Background] Gadducci A, Sartori E, Maggino T, Zola P, Cosio S, Zizioli V, Lapresa M, Piovano E, Landoni F. Pathological response on surgical samples is an independent prognostic variable for patients with Stage Ib2-IIb cervical cancer treated with neoadjuvant chemotherapy and radical hysterectomy: an Italian multicenter retrospective study (CTF Study). Gynecol Oncol. 2013 Dec;131(3):640-4. doi: 10.1016/j.ygyno.2013.09.029. Epub 2013 Oct 3. PMID 24096111
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Rose PG, Bundy BN, Watkins EB, Thigpen JT, Deppe G, Maiman MA, Clarke-Pearson DL, Insalaco S. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1144-53. doi: 10.1056/NEJM199904153401502. PMID 10202165
- [Background] Green JA, Kirwan JM, Tierney JF, Symonds P, Fresco L, Collingwood M, Williams CJ. Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis. Lancet. 2001 Sep 8;358(9284):781-6. doi: 10.1016/S0140-6736(01)05965-7. PMID 11564482
- [Background] Lukka H, Hirte H, Fyles A, Thomas G, Elit L, Johnston M, Fung MF, Browman G; Cancer Care Ontario Practice Guidelines Initiative Gynecology Disease Site Group. Concurrent cisplatin-based chemotherapy plus radiotherapy for cervical cancer--a meta-analysis. Clin Oncol (R Coll Radiol). 2002 Jun;14(3):203-12. doi: 10.1053/clon.2002.0076. PMID 12109823
- [Background] Holden JA. Human deoxyribonucleic acid topoisomerases: molecular targets of anticancer drugs. Ann Clin Lab Sci. 1997 Nov-Dec;27(6):402-12. PMID 9433537
- [Background] Hsiang YH, Hertzberg R, Hecht S, Liu LF. Camptothecin induces protein-linked DNA breaks via mammalian DNA topoisomerase I. J Biol Chem. 1985 Nov 25;260(27):14873-8. PMID 2997227
- [Background] Gupta S, Maheshwari A, Parab P, Mahantshetty U, Hawaldar R, Sastri Chopra S, Kerkar R, Engineer R, Tongaonkar H, Ghosh J, Gulia S, Kumar N, Shylasree TS, Gawade R, Kembhavi Y, Gaikar M, Menon S, Thakur M, Shrivastava S, Badwe R. Neoadjuvant Chemotherapy Followed by Radical Surgery Versus Concomitant Chemotherapy and Radiotherapy in Patients With Stage IB2, IIA, or IIB Squamous Cervical Cancer: A Randomized Controlled Trial. J Clin Oncol. 2018 Jun 1;36(16):1548-1555. doi: 10.1200/JCO.2017.75.9985. Epub 2018 Feb 12. PMID 29432076
- [Background] Neoadjuvant Chemotherapy for Cervical Cancer Meta-Analysis Collaboration (NACCCMA) Collaboration. Neoadjuvant chemotherapy for locally advanced cervix cancer. Cochrane Database Syst Rev. 2004;2004(2):CD001774. doi: 10.1002/14651858.CD001774.pub2. PMID 15106161
- [Background] Wang PH, Chang YH, Yang YH, Chang WH, Huang SY, Lai CR, Juang CM, Chen YJ, Horng HC, Wen KC, Ng HT, Yuan CC, Chao KC, Yen MS. Outcome of patients with bulky IB (>/= 6 cm) cervical squamous cell carcinoma with and without cisplatin-based neoadjuvant chemotherapy. Taiwan J Obstet Gynecol. 2014 Sep;53(3):330-6. doi: 10.1016/j.tjog.2014.05.001. PMID 25286786
- [Background] Li R, Lu ST, Si JG, Liu B, Wang H, Mei YY, Linghu H. Prognostic value of responsiveness of neoadjuvant chemotherapy before surgery for patients with stage IB(2)/IIA(2) cervical cancer. Gynecol Oncol. 2013 Mar;128(3):524-9. doi: 10.1016/j.ygyno.2012.11.006. Epub 2012 Nov 9. PMID 23146686